CLINICAL TRIAL: NCT02433860
Title: Evaluation of the Effectiveness of Pharmacists in Implementing the Smoking Cessation and Reduction in Pregnancy and Treatment (SCRIPT) Protocol
Brief Title: Evaluation of the Effectiveness of Pharmacists in Implementing the SCRIPT Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Providence Medical Research Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A20010724157261
Record Dates: First submitted 2014-10-16; First posted 2015-05-05 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- pregnant nicotine users (Experimental): watch video and tobacco cessation counselling using SCRIPT protocol
  Interventions: Behavioral: pharmacist nicotine cessation counseling using SCRIPT protocol

INTERVENTIONS:
Behavioral: pharmacist nicotine cessation counseling using SCRIPT protocol — Participant will be shown a short DVD "Commit to Quit: During and After Pregnancy. She will be given "a Pregnant Woman's Guide to Quitting" booklet.
  Participant will be asked their nicotine use status and it will be confirmed with a CO meter test and cotinine urine test. Those not consenting to be part of the study will not receive the urinalysis.
  Participant will be advised to quit smoking. The pharmacist will review the Guide with the participant. The participant will receive a phone call around the time of their quit/reduction date. The participant will meet again approximately one week after their quit/reduction date and receive a CO meter test and urine cotinine test.
  At the end of the program pregnant women will answer a follow-up questionnaire. Those women participating in the research study will be given a cotinine urine test at approximately > 36 weeks gestation or at delivery.
  Other Names: Pharmacist counselling using SCRIPT

SUMMARY:
There is a significant need for nicotine cessation programs for pregnant women in Spokane County. SCRIPT has been proven to be an effective method for smoking cessation in pregnant women. This study will evaluate the success of SCRIPT delivered by pharmacists. At the end of the study, the investigators hope to have three questions answered: 1) what is the quit rate of pregnant women in the Spokane area who receive the SCRIPT intervention delivered by pharmacists? 2) How does the quit rate compare to the quit rates of SCRIPT programs delivered by other health care providers as documented in the literature? And 3) Does the SCRIPT intervention have a significant effect on quit rates for pregnant women compared to current Spokane county quit rates? Urine cotinine tests will be used to document smoking status before delivery of the SCRIPT program, approximately one week after quit date and at >36 wks gestation or at delivery for study participants.

DETAILED DESCRIPTION:
1. The goal of this project is to evaluate the success of pharmacists in delivering the SCRIPT smoking cessation program. The research questions that need to be addressed are: i. What is the quit rate of pregnant women in the Spokane area who receive the SCRIPT intervention delivered by a pharmacist? ii. How does this quit rate compare to the quit rates of other SCRIPT programs given by other health care providers (social workers, nurses, etc.)? iii. Does the SCRIPT intervention have a significant effect on quit rates for smoking pregnant women compared to current Spokane county quit rates?

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* nicotine use
* English speaking
* 18 years of age or older

Exclusion Criteria:

* Males due to pregnancy status not applicable

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-01; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
quit rates for nicotine for pregnant women | 2 yrs
  1. The quit rates of pregnant women in this program will be compared to SCRIPT studies to evaluate the effectiveness of pharmacists providing this program.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Taylor, PharmD, Principal Investigator — Providence Holy Family, SHMC and PMP ACC/PHAC
Locations (1):
- Providence Holy Family Hospital Anticoagulation and Pharmacotherapy Clinic, Spokane, Washington, United States